CLINICAL TRIAL: NCT04480229
Title: A Randomized Controlled Study on the Influence of Telenursing Services to the Chemotherapy Treatment of Breast Cancer Patients: The Turkish Case
Brief Title: Telenursing and Breast Cancer: The Turkish Case
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 50687469-1280-2190-14
Record Dates: First submitted 2020-06-03; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer Female
Keywords: telenursing; breast cancer; chemotherapy; symptom management
MeSH Terms: conditions — Breast Neoplasms | interventions — Telenursing; Counseling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): After the first treatment, every week the patients were called and consulted by telenursing. During the next there chemotherapy treatments, Edmonton Symptom Assessment System and General Comfort Questionnaire were filled. The study ended with the fourth cycle chemotherapy. A total of six telephone calls and 3 face-to-face follow-ups were done with each of the intervention group patients. Face-to-face follow-up with patients during chemotherapy treatments lasted for about 20-30 minutes, and patients were evaluated three times in terms of symptom severity and comfort level.
  Interventions: Behavioral: Telenursing and Counseling
- No Intervention: Control Group (No Intervention): During their first treatment the "Patient Identification Form" was filled and they were trained, which is the routine practice of the clinic. Patients were informed about the "Symptom follow-up form", asked to mark the symptoms and signs they experienced due to the disease and treatment in the form between the two chemotherapy treatments and to note when they experienced and how they resolved this symptom. When the patients came to the second treatment, the first follow-up of the patients was done. The investigator filled Edmonton Symptom Assessment System and General Comfort Questionnaire forms via face-to-face interviews. The "Symptom Follow-up Form" given to the patients in the previous chemotherapy treatment was collected and the same new form was given. They were requested to bring this form in their next treatment. The same protocol was followed during the third and fourth chemotherapy treatment

INTERVENTIONS:
Behavioral: Telenursing and Counseling — After the first face-to-face training, counseling on the phone was conducted every week for four cycles of chemotherapy treatment. In total, six counseling sessions and four face-to-face training sessions were conducted for each patient.
  Arms: Intervention Group

SUMMARY:
This study aims to determine the effectiveness of telenursing services on chemotherapy symptoms and comfort levels in patients with breast cancer in Turkey.

DETAILED DESCRIPTION:
This study aims to determine the effectiveness of telenursing services on chemotherapy symptoms and comfort levels in patients with breast cancer in Turkey. The study employs an experimental research methodology with a sample of 96 ambulatory patients (48 experimental, 48 control) who were receiving chemotherapy for breast cancer for the first time in a state hospital. Research data were collected by using "Patient Information Form", "Edmonton Symptom Assessment Scale", "General Comfort Questionnaire, "Symptoms Follow-up Form", and "Telephone Call Form". The experimental group received telenursing service every week until the end of the four-cycle chemotherapy treatment, which started one week after the first treatment. The control group did not receive any intervention. Investigators analyzed data with SPSS 15.0 (Statistical Package for the Social Sciences) with comparative statistical methods of MannWhitney U Test, Chi-Square Test, One Way Analysis of Variance in Repeated Measurements, and Pearson Correlation.

ELIGIBILITY:
Inclusion Criteria:

* is volunteering to participate in the research,
* is 18 years of age or over,
* can communicate in Turkish,
* has Turkish literacy skills,
* has no hearing, vision problems, and mental disability that may hinder communication,
* is female,
* has a diagnosis of breast cancer for the first time in her life and consequently receiving chemotherapy treatment in the same protocols for the first time,
* did not have a different diagnosis of cancer and related chemotherapy treatment.

Exclusion Criteria:

* Having been diagnosed with breast cancer before and received chemotherapy treatment accordingly,
* Having been diagnosed with different cancers before and had chemotherapy treatment related to it,
* Cancer treatment with oral medications,
* Refuse to participate in the study
* Refuse education/counseling
* Not knowing Turkish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Having been diagnosed with breast cancer
Enrollment: 96 (Actual)
Dates: Start 2016-05-06 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
Edmonton Symptom Assessment System | 10 minutes
  This tool is designed to assist in the assessment of symptoms common in cancer patients: pain,fatique, nausea, sadness, anxiety, insomnia, anorexia, wellbeing and shortness of breath, change in skin-nails, mucositis and numbness in hands. The patient circles the most appropriate number to indicate where the symptom is between "0" and "10". "0" is the minimum value, which means there is no change and it is a better outcome for the patient. "10" is the maximum value, means that the symptom level is the highest, which is a worse outcome for the patient.

SECONDARY OUTCOMES:
General Comfort Questionnaire | 10 minutes
  It is used to evaluate the situation of achieving the expected comfort increase result with nursing interventions that provide comfort. The scale, which is a four-point likert type, has a total of 48 items, 24 items are positive and 24 items are negative.
  The lowest value that can be taken is 1 which indicates low comfort and this is a worse outcome. The highest value 4 indicates high comfort, which is a better outcome. The response patterns of the scale, which consists of positive and negative items, are given in mixed form. Accordingly, from positive statements; high score (4p) indicates high comfort, low score (1p) indicates low comfort, while negative items indicate low comfort (1p), high score (4p) low comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Cicek Yagci, Ph.D., Principal Investigator — Istinye University

IPD SHARING:
Plan to Share IPD: No